CLINICAL TRIAL: NCT01825317
Title: Effect of NeuroAD, Combined TMS Stimulation and Cognitive Training, on the Cognitive Function of Mild to Moderate Alzheimer Patients
Brief Title: Effect of NeuroAD on Alzheimer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuronix Ltd (Industry)
Collaborators: company: K The Power (Unknown); Chungnam National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NRX-KOR1
Record Dates: First submitted 2013-04-02; First posted 2013-04-05 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; TMS; NeuroAd; cognitive training; ADAS-Cog
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NeuroAD (Active Comparator): Treatment by the NeuroAD device, real treatment by synchronized TMS+cognitive training
  Interventions: Device: NeuroAD
- Sham NeuroAD (Sham Comparator): Sham TMS+cog, has the same sound and appearance, patients come for the same number of treatments and are exposed to the same procedure.
  Interventions: Device: Sham device

INTERVENTIONS:
Device: NeuroAD — synchronized TMS+COGNITIVE TRAINING
  Other Names: NICE
  Arms: NeuroAD
Device: Sham device — Sham TMS+cog, has the same sound and appearance as the real device, delivers no energy.
  Other Names: Control device
  Arms: Sham NeuroAD

SUMMARY:
Non-invasive stimulation of the brain using magnetic and cognitive stimulation by computer for the treatment of Alzheimer patients.

DETAILED DESCRIPTION:
Synchronized TMS and cognitive training for the treatment of mild to moderate Alzheimer's patients. Treatment is delivered 5 days a week, for 6 weeks, visit is about an hour long.

Evaluation is by neuropsychological evaluation at 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age 60-90 years
2. Patients diagnosed with mild or moderate stage of Alzheimer's Disease, according to the DSM-IV criteria.
3. MMSE score 18 to 26
4. Adas-cog above 17
5. Physically acceptable for the study as confirmed by medical history and exam.
6. Spouse, family member or professional caregiver agree and capable of taking care and be responsible for the participation of the patient in the study (answering questions regarding the patient's condition and assuming responsibility for medication)
7. Agreement to participate in approximately 14 weeks during the study.
8. Normal or corrected to normal ability to see and to hear.
9. Korean as primary language
10. 8th grade education minimum

Exclusion Criteria:

1. CDR 0 or 3
2. Severe agitation;
3. Mental retardation;
4. Patient lacking capacity to consent to study participation
5. Unstable medical condition;
6. Use of benzodiazepines or barbiturates during the study and preceding two weeks;
7. Pharmacological immunosuppression;
8. Participation in a clinical trial with any investigational agent within two weeks prior to study enrollment;
9. History of Epileptic Seizures or Epilepsy;
10. Contraindication for performing MRI scanning;
11. Contraindication for receiving TMS treatment according to a TMS questionnaire;
12. Pregnant women, and women who have the ability to become pregnant unless they are on an acceptable method of contraception during the study.
13. Patients with personal history of any clinically defined neurological disorder, including organic brain disease, epilepsy, stroke, brain lesions, or multiple sclerosis; or personal history of previous neurosurgery or head trauma that resulted in loss of consciousness.
14. Patients with depression, bipolar disorder or psychotic disorders or any other neurological or psychiatric condition (whether now or in the past), which the Investigator finds as interfering with the study
15. Alcoholism or drug addiction as defined by DSM-IV within last 5 years (addicted more than one year and or in remission less than 3 years) or severe sleep deprivation
16. Patients treated with cholinesterase inhibitors, or memantine or Ginko-biloba will be allowed to participate, if the treatment has started at least 6 months previous to recruitment. The patients should keep their dose of medication during the whole trial as prior to study begin.
17. Patients with metal in the head, except the mouth (i.e. cochlear implants, implanted brain stimulators, aneurysm clips)
18. Patients with increased intracranial pressure
19. Cardiac pacemakers
20. Implanted neurostimulators
21. Implanted medication pumps
22. Intracardiac lines
23. Significant heart disease
24. Currently taking medication that lower the seizure threshold
25. Significant sleep deprivation and alcoholism

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
ADAS-Cog | 6 weeks
  Alzheimer's disease assessment scale - cognitive test

CONTACTS AND LOCATIONS:
Locations (1):
- Chungnam national university hospital, Daejeon Geriatric Medical Center, Daejeon, South Korea